CLINICAL TRIAL: NCT06063252
Title: Newly Diagnosed With Inflammatory Arthritis - a Self-management Intervention (NISMA) A Descriptive Randomized Controlled Feasibility Study
Brief Title: Newly Diagnosed With Inflammatory Arthritis - a Self-management Intervention (NISMA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Appel Esbensen, Professor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GlostrupUHN
Record Dates: First submitted 2023-09-12; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Feasibility

STUDY DESIGN:
Intervention Model Description: This feasibility study is designed as a randomized controlled feasibility trial (allocation ratio 1:1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- controlgroup (No Intervention): Usual care
- intervention group (Experimental): receive self-management intervention
  Interventions: Behavioral: NISMA

INTERVENTIONS:
Behavioral: NISMA — The intervention NISMA is a nine-month intervention and consisted of four individual sessions and two group sessions. The theoretical frame is Social Cognitive Theory, along with Acceptance and Commitment Therapy (ACT), to support the enhancement of self-efficacy. It involves four individual face-to-face sessions with a nurse and two group sessions (5-7 patients) with a nurse, an occupational therapist (OT), and a physiotherapist (PT), with the nurse being the facilitator. Every session has a specific topic and, in every session, a person-centered approach was used to address current problems and secure relevance.
  Participants in the control group receive usual care, and the intervention group receives both usual care supplemented with the intervention.
  Arms: intervention group

SUMMARY:
Even though medical treatment has improved within the last 10-15 years, patients with inflammatory arthritis (IA) still experience reduced quality of life, depression, anxiety, changes in family roles, work life, and social relationships. Particularly the newly diagnosed, require regular consultations and available support from health professionals, to be able to handle emotional, social, and physiological challenges.

The hypothesis is that a self-management intervention can improve patients' ability to monitor their arthritis and respond to symptoms, reduce the risk of co-morbidities, and improve adherence. And also, that they can develop cognitive, behavioral, and emotional strategies to manage life with arthritis. There is a lack of disease-specific evidence, in integrated interventions with multiple components targeting patients with a newly diagnosed IA. In a previous study, the investigators developed a self-management intervention, and now wish to test it in a randomized feasibility study.

DETAILED DESCRIPTION:
RATIONALE FOR NISMA PROJECT

The hypothesis is that a self-management intervention can help patients develop behavioral and emotional strategies to manage life with arthritis. There a lack of disease-specific evidence, in integrated interventions with multiple components targeting patients with a newly diagnosed IA. Therefore, the investigators wish to develop a self-management intervention.

Aim

The overall aim of this study is to determine whether a full-scale randomized controlled trial, which aims to increase self-management in patients with newly diagnosed IA, is possible. The investigators wish to identify methodological, clinical, and procedural uncertainties in delivering a self-management intervention. Furthermore, to investigate outcomes related to recruitment, including adherence, retention, accrual rate, characteristics of the sample, and reliable recruitment methods.

Design

This feasibility study is designed as a randomized controlled feasibility trial (allocation ratio 1:1) to assess the proposed method in the definitive RCT.

Overall Setting

The intervention will take place at the Center for Rheumatology and Spine Diseases, Rigshospitalet, Denmark.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons (≥18 years)
* Diagnosed with one of the following diagnoses: Rheumatoid arthritis (ICD10 diagnoses: M05.3, M05.9, M05.8, M06.9), Spondyloarthritis (ICD10 diagnoses: M45.9, M46.1, M46.8, M46.9) or Psoriatic arthritis (ICD10 diagnoses: M073.A, M073.B), within the last 6 months.

Exclusion Criteria:

* Insufficient language skills to discuss the topics in the intervention in Danish
* In chemotherapy treatment for malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Recruitment | Assessed at 3 months
  Recruitment rate will be assessed as the number of patients recruited out of the number of eligiable patients
Retention | Assessed at 9 months
  Retention rate will be assessed as the number of patients who wtihdrew from the study out of the total number of patients.
Adherence | Assessed at 9 months
  Adherence to intervention protocol of the study assessed as the number of sessions attended out of the total number of sessions available

SECONDARY OUTCOMES:
Physical activity measured by the Physical activity and sedentary time questionnaire (FAST) | Assessed at baseline and 9 months
  Physical activity measured by the Physical activity and sedentary time questionnaire (FAST)
Pain intensity measured by the Visual analog scale for pain (VAS) | Assessed at baseline and 9 months
  Pain measured by the Visual analog scale for pain. Score from 0-100. Higher score is more pain.
Functional status measured by the Multi-Dimensional Health Assessment Questionnaire (MD-HAQ) | Assessed at baseline and 9 months
  Functional status measured by the Multi-Dimensional Health Assessment Questionnaire. Score from 0-3. Higher score is more disability.
Fatigue measured by the Bristol Reumatoid Arthritis Fatigue Questionnaire (BRAF) | Assessed at baseline and 9 months
  Fatigue measured by the Bristol Reumatoid Arthritis Fatigue Questionnaire (BRAF). It consists of 20 questions with four responses in four categories: physical fatigue, living with fatigue, cognitive fatigue, and emotional fatigue. Higher score is more fatigue.
Fatigue measured by the visual analog scale for fatigue (VAS-fatigue) | Assessed at baseline and 9 months
  Fatigue measured by the visual analog scale for fatigue (VAS-fatigue). Score from 0-100. Higher score is more fatigue.
Health Literacy was measured by the Health Literacy Questionnaire (HLQ) | Assessed at baseline and 9 months
  Health Literacy was measured by the Health Literacy Questionnaire. Independent scales measuring health literacy on a continuous scale. Scores range between 1 to 4 (for first 5 scales) and 1 to 5 (for scales 6 to 9).
Health related quality of life measured by the EuroQol-5 Dimension (EQ5D) | Assessed at baseline and 9 months
  Quality of life measured by the EuroQol-5 Dimension. measures the patient's self-rated health status. Ranging from -0.624 to 1, higher is better.
Illness perception measured by the Brief Illness Perception Questionnaire (B-IPQ) | Assessed at baseline and 9 months
  Illness perception measured by the Brief Illness Perception Questionnaire. Score from 1-10. Higher is worse.
Self-efficacy measured by the Arthritis specific self-efficacy measurement tool (ASES) | Assessed at baseline and 9 months
  Self-efficacy measured by the Arthritis specific self-efficacy measurement tool. Score from 1-10. Higher score is better
Anxiety and depression measured by the Hospital Anxiety and Depression Scale (HADS) | Assessed at baseline and 9 months
  Anxiety and depression measured by the Hospital Anxiety and Depression Scale. ). HADS is a 14-item questionnaire that assesses levels of anxiety and depression symptoms in medically ill patients in two 7-item sub-scales, one for anxiety (HADS-A) and one for depression (HADS-D). Scores of 8 to 10 suggest the presence of a mood disorder. Scores of 11 or higher indicate the probable presence of a mood disorder. Symptoms of anxiety and depression were defined by scores of 8 or higher.
Disease activity RA measured the Disease Activity Score in 28 joints (DAS28) | Assessed at baseline and 9 months
  Disease activity in rheumatoid arthritis, measured the Disease Activity Score in 28 joints with erythrocyte sedimentation rate. Composite measures, in which multiple aspects of the disease are combined in a total score of the level of disease activity. Higher is worse.
Disease activity SpA measured by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Assessed at baseline and 9 months
  Disease activity in patients with spondyloarthritis, was measured by the Bath Ankylosing Spondylitis Disease Activity Index. The sum score ranges from 0 to 100 with higher values indicating more active disease
Disease activity PsA measured by the the Disease Activity index for PSoriatic Arthritis (DAPSA). | Assessed at baseline and 9 months
  Disease activity in patients wiht psoriatic arthritis, was measured by the Disease Activity index for PSoriatic Arthritis. Composite measures, in which multiple aspects of the disease are combined in a total score of the level of disease activity. Higher is worse.

CONTACTS AND LOCATIONS:
Overall Officials: Bente A Esbensen, Professor, Principal Investigator — Rigshospitalet, Glostrup, Center for Rheumatology and Spine Diseases. COPECARE
Locations (1):
- Luise Holberg Lindgren, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
As this is feasibility outcome data, sharing data i not likely to be relevant

REFERENCES:
- [Derived] Lindgren LH, Thomsen T, Hetland ML, Aadahl M, Kristensen SD, de Thurah A, Esbensen BA. A self-management intervention for newly diagnosed with inflammatory arthritis: a randomized controlled feasibility and fidelity study. Pilot Feasibility Stud. 2025 Feb 11;11(1):15. doi: 10.1186/s40814-025-01601-z. PMID 39934926

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT06063252/Prot_SAP_000.pdf